CLINICAL TRIAL: NCT01545687
Title: A Phase III, Randomized, Double-Blind Study of Lactobacillus Brevis CD2 Lozenges Versus Placebo in the Prevention of Acute Oral Mucositis (OM) in Patients With Head and Neck Cancer Receiving Concurrent Radiotherapy and Chemotherapy
Brief Title: CD2 Lozenges in Preventing Acute Oral Mucositis in Patients With Head and Neck Cancer Receiving Radiotherapy and Chemotherapy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N11C5; NCCTG-N11C5; CDR0000727295 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-00692 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Head and Neck Cancer; Oral Complications of Radiation Therapy; Pain; Weight Changes
Keywords: pain; oral complications of radiation therapy; weight changes; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IVA squamous cell carcinoma of the larynx; stage IVA squamous cell carcinoma of the oropharynx; stage IVA verrucous carcinoma of the larynx; stage IVB squamous cell carcinoma of the larynx; stage IVB squamous cell carcinoma of the oropharynx; stage IVB verrucous carcinoma of the larynx; stage IVC squamous cell carcinoma of the larynx; stage IVC squamous cell carcinoma of the oropharynx; stage IVC verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I verrucous carcinoma of the oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage II verrucous carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IVA squamous cell carcinoma of the lip and oral cavity; stage IVA verrucous carcinoma of the oral cavity; stage IVB squamous cell carcinoma of the lip and oral cavity; stage IVB verrucous carcinoma of the oral cavity; stage IVC squamous cell carcinoma of the lip and oral cavity; stage IVC verrucous carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Pain; Body Weight Changes; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients dissolve in mouth 1 lozenge of Lactobacillus bevis CD2 every 2-3 hours (total of 6 per day) daily during CRT (comprising cisplatin and radiotherapy [RT]) and for 4 weeks after, including weekends.
  Interventions: Dietary Supplement: Lactobacillus brevis CD2 lozenge
- Arm II (Placebo Comparator): Patients dissolve in mouth 1 lozenge of placebo every 2-3 hours (total of 6 per day) daily during CRT and for 4 weeks after, including weekends.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus brevis CD2 lozenge — Dissolved orally
  Arms: Arm I
Other: placebo — Dissolved orally
  Arms: Arm II

SUMMARY:
RATIONALE: Lactobacillus bevis CD2 lozenge may help prevent symptoms of mucositis, or mouth sores, in patients receiving radiation therapy and chemotherapy. This therapy may improve the quality of life of patients with head and neck cancer.

PURPOSE: This phase III trial studies how well Lactobacillus bevis CD2 lozenge prevents oral mucositis in patients with head and neck cancer who are being treated with cisplatin and radiation therapy. These results will be compared to results in patients using placebo lozenges.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether Lactobacillus brevis CD2 lozenges are effective in reducing oral mucositis (OM)-related pain in patients undergoing chemoradiotherapy (CRT) for head and neck squamous cell carcinoma, as measured by the area under the curve (AUC) of Mouth and Throat Soreness (MTS) score (Oral Mucositis Daily Questionnaire [OMDQ] question 2) measured daily during CRT and daily for 4 weeks after completion of CRT.

Secondary

* To assess whether L. brevis CD2 lozenges reduce OM as assessed by the provider using the WHO OM scale, Oral Mucositis Assessment Scale (OMAS), and Common Terminology Criteria Adverse Events (CTCAE).
* To assess whether L. brevis CD2 lozenges reduce the impact of OM on the ability to swallow, drink, eat, talk, and sleep, as assessed by the MTS-Activity Limitations (MTS-AL).
* To assess whether L. brevis CD2 lozenges improve quality of life, as assessed by the Functional Assessment of Cancer Therapy - Head and Neck (FACT-HN).
* To assess whether L. brevis CD2 lozenges reduce opioid requirements.
* To assess whether L. brevis CD2 lozenges improve radiotherapy compliance.
* To assess whether L. brevis CD2 lozenges reduce weight loss and the need for a feeding tube.
* To assess whether L. brevis CD2 lozenges affect disease-free survival (DFS) at 12 months after treatment.
* To evaluate the effect of L. brevis CD2 lozenges on salivary biomarkers, including metabonomic and inflammatory markers, as measured at baseline, week 3 of CRT, and during the last week of CRT. (exploratory)

OUTLINE: This is a multicenter, randomized, placebo-controlled, double-blind study. Patients are stratified according to primary disease site (oral cavity/oropharynx vs nasopharynx vs hypopharynx/larynx), context of chemoradiotherapy (CRT) (definitive vs post-operative), cisplatin schedule (every 3 weeks [100 mg/m^2] vs every week [30-40 mg/m^2]), and use of intensity-modulated radiotherapy (IMRT) (yes vs no). Patients are randomized to 1 of 2 treatment regimens.

* Arm I: Patients dissolve in mouth 1 lozenge of Lactobacillus brevis CD2 every 2-3 hours (total of 6 per day) daily during CRT (comprising cisplatin and radiotherapy [RT]) and for 4 weeks after, including weekends.
* Arm II: Patients dissolve in mouth 1 lozenge of placebo every 2-3 hours (total of 6 per day) daily during CRT and for 4 weeks after, including weekends.

Patients complete questionnaires about their quality of life and pain at baseline and daily during study treatment.

Saliva is collected from some patients before starting RT, during week 3 of RT, and during the last week of RT for NMR-spectroscopic metabolomic analysis and future cytokine analysis.

After completion of study treatment, patients are followed up at 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic proof of squamous cell carcinoma of the oral cavity, oropharynx, nasopharynx, hypopharynx, or larynx
* Planned course of definitive or post-operative radiotherapy (RT) to a total dose of ≥ 60 Gy using 1.8 to 2.0 Gy per fraction
* At least one third of the oral cavity mucosa must be included in the RT fields, as estimated by the treating radiation oncologist
* Planned concurrent administration of cisplatin chemotherapy (either 100 mg/m^2 every 3 weeks or 30-40 mg/m^2 every week)

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0, 1, or 2
* Hemoglobin ≥ 10.0 g/dL
* White blood cell (WBC) ≥ 3,500 x10^9/L
* Absolute neutrophil count (ANC) ≥ 1,500 x10^9/L
* Platelet count ≥ 100,000 x10^9/L
* Willing to abstain from ingestion of yogurt products and/or any product containing probiotics during study drug treatment
* Ability to complete questionnaire(s) by themselves or with assistance
* Willing to provide saliva samples for correlative research purposes (first 50 patients)
* Not pregnant or nursing
* Negative pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential
* Men or women of childbearing potential must employ adequate contraception
* No co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* No current untreated oral candidiasis, oral herpes simplex virus (HSV) infection, or oral mucositis

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No split-course RT planned
* No prior head and neck RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The AUC of the MTS score | Up to 12 months

SECONDARY OUTCOMES:
OM measured by WHO OM scale, OMAS and CTCAE weekly during CRT | Up to 12 months
Impact of OM on the ability to swallow, drink, eat, talk, and sleep, as assessed by the MTS-AL | Up to 12 months
Quality of life as assessed by the FACT-HN | Up to 12 months
Opioid requirement (frequency, morphine equivalent dose) as measured by daily OMDQ | Up to 12 months
DFS at 12 months after treatment | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Miller, MD, Principal Investigator — Mayo Clinic